CLINICAL TRIAL: NCT05872698
Title: Beta-blockers Or Placebo for Primary Prophylaxis of Oesophageal Varices (BOPPP Trial). A Blinded, UK Multi-centre, Clinical Effectiveness and Cost-effectiveness Randomised Controlled Trial.
Brief Title: Beta-blockers or Placebo for Primary Prophylaxis (BOPPP) of Oesophageal Varices Trial.
Acronym: BOPPP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); Cardiff University (Other); Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 255446
Record Dates: First submitted 2021-01-21; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cirrhosis, Liver; Portal Hypertension; Variceal Hemorrhage; Varices, Esophageal
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Esophageal and Gastric Varices | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol (Active Comparator): Oral Carvedilol 6.25 mg to 12.5 mg OD/ or 6.25mg BD (maximum dose 12.5mg)
  Interventions: Drug: Carvedilol
- Placebo (Placebo Comparator): Oral tablet (1 or 2 tablets)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — Carvedilol, sold under the brand name Coreg among others, is a medication used to treat high blood pressure, congestive heart failure, and left ventricular dysfunction in people who are otherwise stable. For high blood pressure, it is generally a second-line treatment. It is taken by mouth.
  Arms: Carvedilol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Research has proven that large varices can be treated with beta-blockers (a type of anti-hypertensive medication) to reduce the pressure in the veins. The management of small varices is still uncertain. This study aims to discover if beta blockers can be used in this setting. We hypothesize that beta blockers will reduce the risk of bleeding from small varices from 20% to 10% over a period of 3 years, resulting in significant cost savings to the NHS from better patient outcomes.

DETAILED DESCRIPTION:
Cirrhosis or liver scarring is an important problem in healthcare in the United Kingdom. 60,000 patients are living with this disease and about 11,000 people every year will die because of it. There are several ways in which patients with this severe form of liver disease become unwell or die and bleeding from the oesophagus or stomach is one. Cirrhosis causes pressure changes inside the abdomen and swelling of veins in the oesophagus (called "varices") which can bleed catastrophically.

We know that when varices are large we need to treat them with medication called beta-blockers to reduce the pressure in the varices. If the varices are small, we are not sure if we need to treat with beta-blockers and this study aims to address this uncertainty. Patients who are recruited to the study with small varices will be randomised to either beta-blockers or a placebo. We will observe them closely for 3 years for bleeding from their varices or other complications of cirrhosis or side effects of taking medication. This is the amount of time needed to observe for bleeding when the varices are small. We will review the patients every 6 months including assessing the varices by a camera test called an endoscopy at the beginning and each year until the study is finished.

During the study patients will be involved with the conduct and management of the research, and we will feedback to recruited patients the results at the end. We will assess the barriers and facilitators of doctors in primary care - such as General Practitioners - in adjusting the dose of the tablets to optimise treatment effects, and assess patients' views on taking part in the trial, and whether the side effects justify the potential benefits of reducing the risk of bleeding. We estimate this risk could be reduced from 20% of patients having significant bleeding to 10% over 3 years.

We will measure the impact of beta-blockers on the overall costs to the NHS of caring for people with cirrhosis during the trial. We will then assess the impact of treatment on both mortality and quality of life using a combined measure, the Quality Adjusted Life-Year (QALY). We will use a mathematical prediction model to estimate the impact of treatment on costs, mortality and quality of life over a patient's lifetime. We will assess whether any increased costs are justified by better outcomes for patients and represent good value for money for the NHS budget.

Finally, we will publish the results of the study in the medical literature and discuss the findings at medical conferences, patient groups and with charities involved in helping patients with cirrhosis such as the British Liver Trust.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Cirrhosis and portal hypertension,
* Small oesophageal varices diagnosed within the last 6 months, defined as ≤5 mm in diameter or varices which completely disappear on moderate insufflation at gastroscopy.
* Not received a beta-blocker in the last week
* Capacity to provide informed consent

Exclusion Criteria:

* Non-cirrhotic portal hypertension
* Medium/large oesophageal varices (current or history [decreasing in size without curative therapy]), defined as >5 mm in diameter
* Gastric (IGV and GOV2), duodenal, rectal varices with or without evidence of recent bleeding.
* Previous variceal haemorrhage
* Previous band ligation or glue injection of oesophageal and/or gastric varices
* Red signs accompanying varices at endoscopy
* Known intolerance to beta blockers
* Contraindications to beta blocker use
* Unable to provide informed consent
* Child Pugh C cirrhosis
* Already receiving a beta-blocker for another reason that cannot be discontinued
* Graft cirrhosis post liver transplantation
* Evidence of active malignancy without curative therapy planned
* Pregnant or lactating women
* Women of child bearing potential not willing to use adequate contraception during the period of IMP dosing
* Patients who have been on a CTIMP within the previous 3 months
* Clinical symptoms consistent with COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Variceal Haemorrhage | 3 years from recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Using a theory-informed approach to explore patient and staff perspectives on factors that influence clinical trial recruitment for patients with cirrhosis and small oesophageal varices — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0263288
- See also: General practitioner perspectives on factors that influence implementation of secondary care-initiated treatment in primary care: Exploring implementation beyond the context of a clinical trial — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0275668